IRB#: 2008540965

# Daily Engagement in Meaningful Activities Professional (DEMA-Pro) intervention for seniors with subjective cognitive decline and living at home

Principal Investigator: Yvonne Lu, PhD, RN, FGSA, FAAN
Professor, Department of Science Nursing Care
Indiana University School of Nursing
600 Barnhill Drive, NU W407
Indianapolis, IN 46202

### **Co-Investigators**

Susan E. Hickman, PhD, Professor, Department of Science Nursing Care Indiana University of School of Nursing

Joan E. Haase, PhD, RN, FAAN
Professor, Department of Science Nursing Care
Indiana University of School of Nursing

Susan M. Perkins, PhD Professor, Biostatistics of Department Indiana University School of Medicine

Pei-Shiun Chang, PhD, RN, MSN, ACNP-BC Assistant Professor, Department of Community Health System Indiana University School of Nursing

Jennifer Ellis, DPT, PhD, GCS Vice President of Research and Business Development, Gentiva Health Services, Inc., d/b/a Kindred at Home.

#### Support Provided by:

NIH, NIA, Protocol Number: AG0700265

NCT#: 04796415

Version Date: 2023 09 12 Page 1 of 1

#### A. SPECIFIC AIMS

Over 4.4 million Americans receive home health services after hospital or rehabilitation facility discharge to improve function, foster independence, promote health-related quality of life and sense of well-being (QoL), and decrease unnecessary hospital or nursing home stays. Among these patients, > 80% are 65 years or older, most manage at least two chronic conditions, and nearly 70% report subjective cognitive decline (SCD).<sup>1-1</sup> SCD is an early clinical sign of Alzheimer's disease and related dementia (ADRD).<sup>2-4</sup> SCD is associated with diminished activity performance, <sup>5-7</sup> poor QoL, <sup>8.9</sup> and other adverse health outcomes (e.g., depressive symptoms).<sup>8,10</sup>

Home health patients with SCD require more time, structure, and guidance to complete tasks and adjust to new skills and environments. Without support, they often lose their sense of control, have fewer personal choices, <sup>11</sup> and disengage from *meaningful activities*. <sup>12,13</sup> Meaningful activities are self-identified activities based on the individual's previous life experiences, sense of intentionality, and goals to remain involved in desired activities and personal relationships. <sup>14,15</sup> In older adults, engagement in meaningful activities is associated with better physical and mental health, QoL, reduced risk of cognitive decline and mortality. <sup>14,16,17</sup> Poor engagement in meaningful activities results in rapid patient decline <sup>18</sup> that may otherwise be preventable. For those with SCD who are at risk of declining and progressing to preclinical ADRD, <sup>19</sup> new care delivery models that promote engagement in meaningful activities to enhance patient outcomes are needed. Because informal caregivers are usually unprepared, lack confidence in their new caregiver role, and have difficulty providing support, <sup>1,20</sup> it is vitally important to include these caregivers in new care delivery models.

We propose a new home health care delivery model in partnership with Kindred at Home (KAH) Gentiva Health Services, a division of Humana that encompasses 400 sites across 40 states. Our proposed telephone-delivered care model, Daily Engagement in Meaningful Activities-Professional (DEMA-Pro) is a *Positive Health* intervention<sup>21</sup> that is strengths-based, family-centered, and tailored to patient/caregiver goals and values. DEMA-Pro addresses the core problem of diminished engagement in meaningful activities among SCD patients at home by: 1) coaching patient-caregiver dyads to problem-solve; 2) teaching the dyads self-management and communication skills; and 3) enhancing naturally occurring patient-caregiver interactions necessary to accomplish self-identified, mutually agreed upon goals. DEMA-Pro builds on five preliminary studies of the DEMA intervention<sup>22-28</sup> that demonstrated high feasibility, acceptability, and positive preliminary effects on health outcomes (physical function, mood, and QoL).<sup>27,28</sup> DEMA-Pro will be refined for delivery by home health services staff to patients with SCD and their informal caregivers.

The purpose of this R61/R33 grant proposal is to conduct a pragmatic cluster randomized controlled trial (RCT) of DEMA-Pro to improve outcomes in home health service patients with SCD. In the R61 phase, we will establish the organizational structure and processes and pilot test DEMA-Pro in 4 KAH home health service facilities. In the R33 phase we will conduct a full pragmatic RCT in 40 KAH facilities to compare DEMA-Pro to usual care. In accordance with pragmatic trial principles, we will primarily use existing data sources including electronic Medicare OASIS (Outcome and Assessment Information Set) data to characterize the cohort and measure outcomes. **R61 and R33 Specific aims** are:

#### R61 Phase (12 months)

**Aim 1**. Establish the organizational infrastructure and programmatic processes needed to conduct a pragmatic cluster-randomized control trial of the DEMA-Pro intervention versus usual care. A Steering Committee will lead the project and coordinate the activities of 3 Work Groups: Regulatory and Operations; DEMA-Pro Intervention Protocol; and Data Management and Analysis.

**Aim 2.** Pilot test the DEMA-Pro training protocol in 4 KAH North Region locations and refine as indicated.

### R33 Phase (48 months).

Forty KAH home health services sites will be randomized to DEMA-Pro or usual care. DEMA-Pro site home health services staff will be trained as DEMA-Pro coaches who will work with home health service leaders to: (1) consolidate home health services DEMA-Pro procedures; (2) train and educate staff; and (3) facilitate DEMA-Pro coaching with patients and their family caregivers. The implementation period will be 18 months and all enrolled patients will be followed for 12 months.

<u>Aim 3.</u> Compare outcomes of DEMA-Pro to Usual Care over 12 months. <u>Hypotheses (H).</u> Compared to usual care, DEMA-Pro patients will have: H 3.1(primary) higher physical function; H 3.2 higher overall quality of life (i.e. Sense of well-being) (QoL); H 3.3 lower depression, and, H 3.4. lower rates of transfers to nursing home per 1000 person days. **Impact:** By valuing and fostering a positive health model of care, an efficacious DEMA-Pro has potential to facilitate a paradigm shift in how elderly patients in the USA are cared for at home. **B. SIGNIFICANCE: R61/R33** 

SCD provides a critical window of time to provide early interventions to slow the onset of dementia and improve negative outcomes. SCD patients and their caregivers need early, supportive interventions from home health services staff to slow functional decline and improve health outcomes. While there are no proven cures or treatments for Alzheimer's disease and related dementia (ADRD), there is strong evidence that combining four or five healthy lifestyle behaviors (i.e., heathy diet, regular exercise, cognitive stimulation, non-smoking, social activity) decreases risk of AD, compared to having none or only one of the five behaviors. However, two of these behaviors, cognitive stimulation and exercise, are less likely to be meaningful enough be sustained by older persons' over time or foster engagement in additional activities. Very few interventions focus on SCD patients and their caregiver in home health services settings. The Institute of Medicine recommended research on active engagement of both patients and their caregivers as a fundamental feature of successful interventions, but few dyadic interventions are developed, tested, or evaluated in the home health setting. Tailored positive health interventions for SCD patients living at home are sorely needed, and opportunities to intervene before progression to moderate/advanced dementia are few.

Patient-driven care and meaningful activity engagement are critical components of home health services. Sustained engagement in meaningful activities is essential for patient QoL. 15.62 Home health services *should* optimize the abilities of patients with SCD and QoL, through engagement in meaningful activity. 63 Unfortunately, healthcare teams often lack important information regarding patient goals, values, and preferences necessary to develop appropriate plans of care. Also, very few supportive care interventions focus on SCD patient-

informal caregiver dyads and none promote reengagement in preferred meaningful activities to maximize QoL, preserve activity performance, prolong independence, and delay institutionalization. Current SCD interventions are rarely tailored to patient preferences, do not involve caregivers, 55,58 and are not easily integrated into the well-established, daily routines. Dyadic engagement in self-selected meaningful activities may be an efficient means to: 1) improve patient and caregiver confidence to manage patient's daily challenges, 15,64 2) promote long-term engagement in meaningful activities; 14,18,65 3) foster feelings of pleasure, connectedness, identity, 14,64 autonomy, and goal directedness; 14,26-28 and, 4) enhance patient activity performance over time 14,15—all of which are important to maintain patient abilities. **Mutual engagement in daily meaningful activities can enhance the patient-caregiver relationships**, 15,66 and enhance both patient and caregiver QoL.25

The Daily Engagement in Meaningful Activities (DEMA) intervention is a practical, promising solution to improve QoL for home health service patients with SCD and reduce caregiver burden. To ensure effective health promotion and quality engagement, DEMA fosters full patient engagement, with caregiver support, to identify meaningful activities, assess capacity, problem-solve barriers, and establish routines for engagement. Our previous studies found prevention of patient disengagement requires a structured, goal-setting approach to foster continued or renewed engagement in diverse meaningful activities. DEMA's highly person-centered approach to activity engagement begins with the patient identifying valued activities and addressing the individual's unique barriers to engagement. Meaningful activity engagement promotes patient and caregiver life satisfaction by coaching the dyad on problem-solving, self-management, active listening, and communication skills, and by enhancing naturally occurring patient/caregiver interactions to accomplish self-identified and mutually agreed upon goals.<sup>26,27,49</sup>

Regardless of whether patients progress to ADRD, remain stable, or improve, <sup>67</sup> patients and caregivers can benefit from DEMA-Pro. This R61 will lead to an R33 pragmatic trial by: 1) creating the organizational structure in the R61 (pilot) phase to be used in the R33 phase; 2) recruiting participants across 4 home health service locations; 3) adapting the DEMA training protocol in collaboration with the KAH professional team to create DEMA-Pro; and, 4) using blended learning modules (i.e. electronic and in-person delivery).

**IMPACT**. SCD is a risk factor for developing Alzheimer disease (AD). Over five million Americans had dementia in 2019, with projections of 7.1 million by 2025. Innovative interventions to address the growing demands for high quality care in this population, and foster both health-related quality of life, quality of life as overall sense of well-being are needed. The interprofessional, telephone delivered DEMA-Pro program, aimed to improve quality of care and patient health outcomes, offers an efficient, cost-efficient care model.

#### C. INNOVATION: R61/R33

<u>DEMA</u> is the first telephone-delivered intervention for patients with SCD and caregivers with demonstrated high feasibility, acceptability, and positive preliminary effects on health outcomes (physical function, mood, and QoL).<sup>27,28</sup> DEMA is primarily telephone delivered (1 in-person and 5 telephone session) and 5 preliminary studies demonstrated very high feasibility: 98% participant consent and 94% completion,<sup>27</sup> indicating *unusually high* patient and caregiver acceptance, minimal burden, and intervention value, compared to other studies of older adults with cognitive impairment (completion rates 60 to 78%).<sup>69-72</sup> DEMA participants reported high satisfaction with the intervener information provided over time. Group comparisons, DEMA mean scores were significantly higher for overall satisfaction subscale:

usefulness (p=.025) and ease of use (p=.038).<sup>28</sup> Participant's post intervention interviews support the helpfulness of DEMA (e.g., Patient: "(DEMA) let me know I'm not the only one...There are things that you can do...to resolve or make them not as big of a problem ... the daily logs showed I was doing much more than I believed." Caregiver: "A program like this is extremely important. If nobody pays any attention...there's no improvement, there's nothing. Most helpful [was] understanding the challenges of memory impairment, learning and practicing a variety of coping skills, and realizing I need to reach out for help without guilt feeling".<sup>28</sup>

The DEMA-Pro intervention will be the first to address the engagement constraints of older persons with SCD using a Positive Health approach to *foster sustainable* engagement in meaningful activities that are based on the shared values and priorities of both patients' and caregivers'. There is emerging evidence that regular, personalized, and self-identified engagement in any meaningful activities can improve quality of life, depressive symptoms, anxiety, and dyad communication. 14,15,65,73,74 The DEMA-Pro Program is: 1) tailored to patients' activity priorities and functional abilities; 2) flexible in activity selection (e.g. one long-term or several short-term activities); 3) collaborative between the patient and caregiver in developing and executing the personalized meaningful activity plan; and; 4) relevant and tailored to patient/caregiver's priority needs for written information related to the 6 priority topics identified and evaluated by focus groups. 27,28,30,31

DEMA-Pro will be the first large-scale pragmatic RCT to evaluate a telephone intervention embedded in existing home health services teams' care for patients with SCD and their family caregivers (Aims 1-3). DEMA-Pro delivery within a pragmatic RCT increases likelihood of success and sustainability. Advantages of this pragmatic trial approach include: 1) coordinated training; 2) DEMA-Pro delivery by dedicated KAH Call Center coaches in collaboration with home health services providers in the field; and, 3) flexible incorporation of DEMA-Pro into home health services policies and procedures. For example, KAH home health service teams will train the KAH Call Center care coordinators to deliver DEMA-Pro and create DEMA-Pro care plans to be implemented by clinical staff in the field with the aim to enhance patient and caregiver engagement in self-selected meaningful activities in home settings. The field staff will be meeting regularly to support the patients in reaching their goals based on the plan created by the coach in the call center. DEMA-Pro will also be integrated into the home health services culture and existing administrative structures, which drives change in home health services settings. For example, the DEMA-Pro Coach will have accountability to their supervisors for their activities as part of their position. Internally generated benchmarking will increase willingness to devote time and resources by elevating the profile of this important staff function.

**DEMA** is efficiently delivered in home settings and DEMA-Pro will leverage DEMA's lessons-learned through delivery as a demonstration project in one of the largest home health services companies in the USA (Aim 1). The DEMA-Pro Program capitalizes on our team's experiences delivering a highly person-centered approach to activity engagement based on patient-identified valued activities and addressing the individual's unique barriers to engagement. Meaningful activity engagement fosters better patient physical function and quality of life (sense of well-being) by coaching dyad problem-solving, self-management, active listening, communication skills, and by enhancing the naturally occurring patient/caregiver interactions to accomplish self-identified and mutually agreed upon goals. Regardless of whether patients with SCD progress to AD, remain stable, or improve, patients and caregivers can benefit from DEMA-Pro.

Our proposed study combines multiple sources of data to comprehensively evaluate quality and effectiveness of DEMA-Pro when delivered through home healthcare services (Aim 3). Use of multiple existing databases to evaluate the quality of home health services for patients with SCD is extraordinarily difficult. Our use of combined data from the Medicare OASIS electronic health record and from KAH's Electronic DEMA-Pro care plan is innovative and will enable us to meaningfully evaluate DEMA-Pro's influence on home healthcare quality of care.

#### D. APPROACH: R61/R33

Following the instruction and requirements provided in RFA-18-585, this section includes description of: (1) preliminary studies relevant to the R61/R33 phases; (2) a conceptual model; (3) detailed methods to assess R61 milestones prior to R33 phase; (4) R33 milestones; and, (5) Potential problems and alternative solutions.

D.1. Preliminary Studies. Our combined expertise is necessary for the success of this DEMA-Pro pragmatic pilot project. PI (Lu) has developed and led a DEMA program of research focused on positive health, strength-based and family-center interventions to improve the meaningful activities, physical function, and quality of life of older adults with cognitive impairment and their family caregivers in past 15 years. Dr. Hickman (Co-I) has significant experience with implementing and evaluating evidence-based interventions for older adults in real world clinical settings, including serving as an 8-year Co-I on a Centers for Medicare and Medicaid Services funded demonstration project in which they are implementing systematic advance care planning in 19 nursing facilities. Dr Haase (Co-I) has extensive experience developing psychosocial behavioral interventions and evaluating them in multi-site randomized clinical trial. Dr. Ellis (Co-I), Vice-President, Research and Business Development, Kindred at Home, has extensive experiences coordinating and leading efforts to guide large-scale implementation of healthcare delivery innovation via translation of evidence to real-world application in large, complex and highly-matrixed healthcare delivery organizations for over 15 years. Dr. Perkins (Co-I) is has extensive statistical experience, serving as biostatistician or Co-Investigator on 33 funded studies (including NIH). Dr. Jones (Consultant), has successful experiences with recruitment and stakeholder engagement in home healthcare setting and recently conducting improving care coordination between clinicians to optimize care transitions to home health care (AHRQ, K08HS024569).

**DEMA-Pro** is adapted from DEMA. DEMA was developed using NIH's Stage Model for Behavioral Intervention Development<sub>95</sub> across five preliminary studies (T32NR007066, P30AG10133-pilot study, K01NR010854, R21NR013755); <sup>23-28</sup> all five studies were consistently focused on patients' and caregivers' self-identified needs and experiences. The studies demonstrated DEMA's high feasibility and acceptability in home settings. Compared to other studies of older adults with cognitive impairment in which completion rates ranged from 60% to 78%, <sup>69-72</sup> we had a 98% consent rate and a 94% completion rate, indicating unusually high acceptance, minimal burden, and high intervention value.<sup>27,28</sup> This pilot offers the unique opportunities to adapt DEMA to the home health service setting, delivered by centralized health care professionals and with evaluation support.

Indiana University & Kindred at Home, Gentiva Health Services academic/corporate research partnership. Kindred at Home (KAH) is one of the largest home health services in the United States (> 400 sites in 40 states). To Dr. Lu (PI) and KAH Vice President Dr. Ellis have collaborated since 2015 on preliminary studies of DEMA, which yielded 2 publications, 28,76 1 manuscript in progress, and 2 poster presentations at national and international conferences. Tr.78

In her role as Vice President of Research and Business Development, Dr. Ellis facilitated a formal memorandum of understanding (MOU) between IU School of Nursing and KAH to collaborate on research and share data (Data Use Agreement No.1153529). This call for pilot proposals is timely, since Drs. Lu, Ellis, and the Chief Officers of KAH had already started exploring adapting the DEMA program for use in the home health services settings—this funding mechanism provides the ideal opportunity to both adapt and rigorously evaluate the implementation of DEMA for dissemination both within and potentially beyond KAH. (See attached of **Letter of Support**).

Team experience conducting pragmatic RCTs with Alzheimer's patient, caregivers, and healthcare providers. As an MPI on a R21/R33 APPROACHES pragmatic clinical trial to implement an advance care planning intervention for persons with ADRD in nursing facilities (R21 AG057463; R33 AG057463), Dr. Hickman established the infrastructure to conduct a pragmatic RCT, developed a training plan, collaborated with corporate partners to adapt intervention protocols, and is using existing federally collected data (Claims, MDS) along with electronic health record (EHR) data to evaluate target outcomes.



**Conceptual Framework (see Figure 1.)** A modified Donabedian<sup>79</sup> approach to quality measurement guides this study. The 4 elements of the model are: 1) context, 2) process, 3) systems of care, and 4) outcomes. In this framework, DEMA-Pro is a process that is influenced by context (e.g. patients/caregiver characteristics) and systems of care (e.g. the KAH home health services sites), to improve intermediate (e.g. meaningful activity engagement) and longer-term outcomes (e.g. physical function, QoL, and reduced depression, hospitalization, emergency visit, and/or transfer to nursing home rates).

### D.3. APPROACH R61 Pilot Phase

<u>Activities to Support Aim 1</u>: Establish the organizational infrastructure and programmatic processes needed to conduct a pragmatic cluster-randomized control trial of the DEMA-Pro intervention versus usual care.

- **D.3.1. Establish Memorandum of Agreement.** PI Lu and Dr. Ellis will work with the IU Office of Research Administration and KAH. Electronic copies of the signed MOU will be securely filed in the IUPUI research office and sent to the NIA Agency. In the R61 phase, patient recruitment and assessment will be done by Assessment Associates at 4 KAH sites; DEMA-Pro will be delivered by protocol-trained personnel at KAH's Centralized Call Center and the resulting DEMA-Pro care plans will be implemented by site clinical staff.
- **D.3.2. Establish Organizational Structure.** As PI, Dr. Lu will oversee all aspects of project development, implementation, and analysis including human resources, NIH/NIA Program Officer communication, and budgetary decisions. **Figure 2** depicts the organizational structure for both the R61 and R33 phases.



**Committee**. Responsibilities are: 1) project oversight, including collaboration between IU and KAH partners, coordinating workgroup tasks, and achieving project milestones, including primary oversight of the pilot pragmatic phase, and transition to the R33 phase; 2) monitoring KAH electronic and Medicare OASIS data to ensure quality of all DEMA-Pro outcome data.

Regulatory and Operations Workgroup. Responsibilities are: 1) obtain a signed MOU from KAH, Gentiva Health Services for the DEMA-Pro trial; 2) follow the signed data use agreements from KAH to ensure access to electronic health record OASIS data<sup>80</sup> and other relevant data; 3) oversee human subjects' protection, obtaining Indiana University Institutional Review Board of Record (IRB of record) approval, and requesting an informed consent waiver for patients and caregivers; 4) coordinate data safety monitoring board (DSMB), convening meetings and supporting data safety and monitoring reporting.

**DEMA-Pro Intervention Protocol Workgroup**. Responsibilities include adapting the DEMA protocol, training protocol and toolkits according to KAH's blended learning modules for use as DEMA-Pro to be implemented as a new KAH initiative. In collaboration with KAH Gentiva Health Servcies, relevant corporate policies will be reviewed and potentially modified or created to support the roll-out of this new initiative. The Chief Officer (O'Sullivan) of KAH Home Health Services confirmed her willingness to make modifications to policies and procedures to support DEMA-Pro. DEMA training and intervention protocols and toolkits will be revised as DEMA-Pro to assure the home health services call-center care coordinators delivering DEMA-Pro coach are able to follow the intervention protocol. DEMA-Pro will be refined based on collaboration and consensus, national standards, and existing research evidence.

Separate meetings will be conducted with each KAH site (n=4) recruiting participants and with home health services corporate leadership to discuss opportunities and potential barriers to implementing DEMA-Pro at the site. DEMA-Pro will be refined based on this feedback and further reviewed with representatives from all 4 sites. Based on feedback, DEMA-Pro materials will be refined and finalized for KAH training and delivery.

A minimum of three KAH call-center care coordinators will be designated DEMA-Pro coaches will receive in-depth training (approximately 8 hours) and hard-copies of the protocol, sample template workflows, educational handouts (i.e. Self-Management Toolkits), and tips for navigating common barriers. Training will include specific information about the principles of problem-solving for patients with SCD and their family caregivers. Core expectations for DEMA-Pro include education provided to KAH staff with dedicated time to coordinate and facilitate discussions with SCD patients and their caregivers. Based on our previous DEMA study personnel training, DEMA-Pro delivery to SCD patients and caregivers requires 60 minutes for each of the six weekly calls. Dedicated time and flexible schedules are important for the DEMA-

Pro coach to facilitate conversations with SDC patients and their caregivers. Consistent with the principles of a pragmatic trial, instructions for the DEMA-Pro coach will be highly flexible.<sup>81</sup>

Per standard operating procedures, a Clinical Assessment Associate at each KAH site will collect and enter data into the electronic health record-OASIS. This Associate will receive one-hour of training to ensure data collection fidelity at both admission and discharge data collection times. In addition, a 20 minutes online video will be provided to other home health services field-based staff to orient them to the goals and processes of DEMA-Pro and to support their use of the DEMA-Pro care plans with patients in the home setting. These KAH home health services field-based staff include registered nurses, physical therapists, occupational therapists, and social workers. The DEMA-PRO coach communicate with to the field-based staff through electronic DEMA-Pro care plan. Adaptations to the DEMA-Pro Self-Management Toolkit, workflows, and educational materials will be made following the pilot.

Data Management and Analysis Workgroup. This group is responsible for obtaining and monitoring all KAH facility and patient data. Based on power calculations, we need 40 KAH home health services locations (20 intervention and 20 control sites, 25 patients/per site; a total of 1000 patients) for the R33 clinical trial phase. This workgroup is responsible for: 1) data management required to link data sources in preparation for analysis and for the actual analysis; 2) data collection protocol and data transfer processes; and 3) the REDCap data management system for the QoL outcome. In Month 2, initial data collection protocol and process for integrating KAH electronic data sources will be tested to determine if any data revisions are necessary. To assess completeness and accuracy of , an electronic health record-OASIS dataset tool, will be compared to the KAH hospitalization rate, or/and transfer to nursing home rate to determine whether the process of merging was accurate. For example, validity checks will be performed to insure all participant hospitalizations and transfers to nursing homes are captured. This also will provide an opportunity to pilot test data cleaning procedures and initial analytic capabilities of the merged data set.

# <u>Activities to Support Aim 2</u>, Pilot test the DEMA-Pro training protocol in 4 KAH North Region sites and refine as indicated.

**D.3.3.1 Pilot Study Setting.** KAH, Gentiva Health Services is a subsidiary of Humana and annually provides home health services to >500,000 patients at > than 400 United States sites in over 40 states. KAH employs teams of clinicians who provide in-home visits with the support of clinicians who provide support and monitoring by phone from the KAH-wide call-center. Call-center care coordinators will deliver DEMA-Pro intervention via telephone. The expected outcome of <u>each</u> session is a DEMA-Pro plan/revised plan for engagement in meaningful activity over the next week. The home health field-base staff will review the electronic weekly DEMA-Pro care plan with participants and support patient and caregiver engagement in meaningful activity according to latest plan. See **Table 1** for R61 (pilot) phase potential number of staff and admissions rates at potential sites.

Table 1. R61 KAH North Region Sites and Numbers of Site Staff and Patient Admissions in 2018

| Location | Number of Staff* | 2018 Patient Admissions |
|-----------------------------|------------------|-------------------------|
| North Region Location No. 1 | 20 | 659 |
| North Region Location No. 2 | 20 | 554 |
| North Region Location No. 3 | 38 | 900 |

| North Region Location No. 4 | 18 | 347 |
|-----------------------------|----------|-------------------------|
| Total | 96 Staff | 2460 Patient Admissions |

<sup>\*</sup>Staff includes nurses, physical therapists, occupational therapists, and speech therapists. **D.3.3.2. R61 Study Population.** There are two study populations.

- 1) <u>KAH staff</u> including call-center care coordinators, clinical assessment associates, field-based therapists, and clinical operational coordinator;
- 2) <u>Home health service patients</u> aged  $\geq$  60 years with SCD, with an OASIS- Cognition Function Subscale Score of 1 or 2 (0 = alert/oriented, able to focus and shift attention, comprehends and recalls task directions independently; 1 = Requires prompting [cuing, repetition, reminders) only under stressful or unfamiliar conditions; 2 = Requires assistance and some direction in specific situations [for example, on all tasks involving shifting of attention] or consistently requires low stimulus environment due to distractibility; 3 = Requires considerable assistance in routine situations. Is not alert and oriented or is unable to shift attention and recall directions more than half the time; 4 = Totally dependent due to disturbances such as constant disorientation, coma, persistent vegetative state, or delirium.

#### D.3.3.3. R61 Data Elements.

Data elements include home health services characteristics (size, rural/urban location), patient characteristics (demographics, cognitive status, and functional status), patient outcomes, and feasibility of DEMA-Pro training and delivery. Consistent with the principle of pragmatic clinical trials, 82.83 primarily existing data will be used to evaluate outcomes. See **Table 2** for Outcomes, Measures and Electronic Data Sources.

The primary study outcome is physical function, assessed using existing OASIS Activity Daily Living and Instrumental Activity Daily Living (ADL/IADLs) subscales. So Secondary outcomes are QoL, depression, the rates of hospitalization, emergency room admission, and transfers to a nursing home. We will use OASIS to assess rates of hospitalization, emergency room visits, and transfer to nursing home. OQL (Sense of Well-being) will be measured with the NIH Toolbox-Psychological Well-being Short-From. Depression will be assessed using the OASIS-PHQ-2 subscale. DEMA-Pro training acceptability, delivery confidence, and ability to meet goals will be assessed using of the existing KAH online learning management system and tools and will be analyzed by the Data Management Workgroup.

Table 2. R61 Data Elements: Patient, Staff, and Outcomes

| Patient Data | Measure(s) | OASIS-D <sup>a</sup> | Other<br>Sources |
|---|---|---|---|
| Demographics | Patient Characteristics | M0010, M0014, M0020,<br>M0030, M0050, M0066,<br>M0069, M0140, M0100,<br>M1000, M1021; M1023,<br>M1028, M1033, M1100,<br>M1200 | |
| Cognitive status | Cognitive Function | M1700 | |
| DEMA-Pro care plan | DEMA-Pro Care Plan and Daily<br>Meaningful Activity Log | | KAH -DEMA-<br>Pro care<br>plan ♭ |
| Staff Data | | | |
| Staff Experiences of DEMA-<br>Pro training and delivery | Feasibility and Acceptability of DEMA-<br>Pro training and delivery survey | | KAH LMS∘ |
| Outcomes Data | | | |

| Physical Function,<br>(Primary Outcome) | Activities of Daily Living/Instructive<br>Activities of Daily Living | M1800, M1819, M1820,<br>MM1830, M1840,<br>M1845, M1850, M1870, | |
|---|---|---|---|
| QoL (Sense of Well-<br>Being) | NIH ToolBox: Psychosocial Well-being-<br>Short-Form | | REDCap |
| Depression | PHQ-2 | M1730 | |
| Hospitalization Rate | Frequency of rehospitalization rate | M2410 | |
| Number, Types of ER visits | Frequency unplanned urgent care or hospital ER care | M2301, M2041 | |
| Nursing Home Transfers | Frequency of transfers to nursing home care | M2410 | |

<sup>&</sup>lt;sup>a</sup>OASIS-D = Outcome and Assessment Information Set Data; <sup>b</sup>KAH electronic DEMA-Pro Care Plan; <sup>c</sup>KAH LMS = Kindred at Home Learning Management Systems.

## **D.3.3.4. R61 Data Collection Protocol.** <u>Patient data</u> will be obtained by a KAH Clinical Assessment

Associate at start of care date, date of any re-admission, and discharge date, using existing KAH electronic data sources including electronic health record-OASIS, Electronic DEMA-Pro Care Plan, learning management system (LMS) and REDCap.

Staff data related to orientation, training, DEMA-Pro delivery and data collection will be obtained from DEMA-Pro coaches, Clinical Assessment Associates, and home health field-based staff. The KAH call-center Care Coordinator will complete the Weekly Activity Engagement Form through the electronic KAH E DEMA-Pro care plan data are used by KAH to identify quality improvement opportunities, evaluate the quality of service provided and guide operational decisions. Items specific to DEMA-Pro outcome s (i.e., QoL) will be added to the KAH home health services REDCap system. KAH staff perception of feasibility of and satisfaction with DEMA-Pro training and delivery survey questions will be added to and entered into KAH LMS.

To establish acceptability of the blended learning modules to train home health providers to deliver DEMA-Pro, the Intervention Protocol Workgroup will: 1) review corporate policies relevant to DEMA-Pro implementation at KAH; 2) adapt the DEMA intervention protocol, training protocol, and Self-Management Toolkit, into blended learning modules and training materials; 3) develop the 15-minute orientation video for KAH home health services field-based staff in Month 4, at the KAH Education/Training Center in Atlanta, and 4) work with KAH clinical operational coordinators to ensure the training protocols are aligned with KAH policies. The Data Management and Analysis Workgroup will: 1) integrate the feasibility and satisfaction survey questions of DEMA-Pro training and delivery into the KAH online system; 2) ensure the KAH trained staff (i.e. call-center care coordinators, clinical assessment associates, home health service field-based staff) complete the feasibility DEMA-Pro training survey after training sessions and the satisfaction survey (within 48 hours of completing training session) in the KAH online system as following the KAH policies; 3) complete the survey data analysis; and 4) provide the results to the steering committee and the funding agency quarterly. PI Lu and the project manager will work with the DEMA-Pro intervention protocol work group to train KAH staff using the modified training protocol, developed blended teaching modules, and training materials.

To assess feasibility of the DEMA protocol as delivered by trained call-center care coordinators, PI Lu will work with the Project Manager and the DEMA-Pro Intervention Protocol Workgroup to

ensure trained KAH call-center care coordinators can follow the DEMA-Pro protocol and deliver the sessions through telephone.

To assess acceptability and quality of study data using the electronic health record- OASIS data collection tool, KAH Electronic DEMA-Pro care plan, and other measures (e.g., QoL), Dr Lu, the (TBD) Project Manager, and the Data Management and Analysis Workgroup will: 1) extract necessary home health services OASIS administrative data, and generate preliminary statistics; 2) access the acceptability and quality of study specific data such as electronic health record from the OASIS data set, the KAH electronic DEMA-Pro care plan, the REDCap Data (e.g. QoL), and KAH online learning management system (e.g. feasibility of DEMA-Pro training and delivery survey data).

**D.3.3.5. R61 Intervention Monitoring** data will be obtained and monitored within the DEMA-Pro REDCap and KAH electronic DEMA-Pro care plan data bases, as modified by the Steering Committee. These modifications are necessary both to monitor the use of the intervention and to support best clinical practice. A goal will be to minimize the burden on staff and maximize the integration of monitoring into existing clinical systems, consistent with the goals of a pragmatic clinical trial. Specifically, the KAH electronic DEMA-Pro care plan will capture: 1) When a DEMA-Pro is held; 2) what is discussed (check box), 3) who are involved; 4) length of discussion, and 5) outcomes (e.g. code status documentation "Weekly Activity Engagement"). The DEMA-Pro coach will be given an assignment list of 5 home health patients with SCD with a total of 20 telephone session monthly approach; the project staff will work with the DEMA-Pro coach and the KAH Clinical Operations Coordinator to determine procedures for generating this monthly assignment list. If a patient or family caregiver is approached by phone, but declines or does not engage (e.g., passive refusal) after three phone call attempts, the DEMA-Pro coach will document this outcome in the electronic DEMA-Pro care plan.

**D.3.3.6. R61 Phase Data Analysis. Analytic Plan.** Aim 1 will not require quantitative analysis. The data collected for Aim 2 will be analyzed with descriptive methods. Item responses will be tabulated and scale scores for acceptability and feasibility summarized by means and standard deviations (or medians and 25<sup>th</sup> and 75<sup>th</sup> percentiles if the data is skewed). Acceptability, feasibility, and satisfaction data will be summarized separately for DEMA-Pro coaches, clinical assessment associates, and home health field-based staff. With respect to patient outcomes, our primary goals are to examine the data collected from the EHR for quality and ensure it can be captured and merged efficiently and appropriately. We will also generate descriptive statistics for all patient outcomes collected through the EHR to help us to identify any data issues, such as missing data patterns, that could influence the implementation of the pragmatic RCT. Cronbach's alpha will be calculated for multi-items scales.

**D.3.3.7. R61Go/No-Go Criteria, Milestones and Timeline.** The Go/No-Go Criteria are established per the RFA guidance to identify the milestones that must be achieved during the R61 phase to qualify for the transition from the R61 to the R33 phase. The R61 Go/No-Go criteria are: 1) Establish partnerships with the KAH home health services as demonstrated by executed memoranda of understanding and data use agreements; 2) Obtain access to necessary administrative data including OASIS, KAH electronic DEMA-Pro care plan, REDCap and KAH LMS; 3) Produce the DEMA-Pro protocol; and 4) Pilot test the DEMA-Pro Program and generate preliminary feasibility data. Milestones and the study timeline are in **Table 3.** 

Table 3. R61 (Pilot) Milestones and Timeline.

| Milestones | Months: | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Start-UP: hire staff, obtain IRB approvals; establish goal timelines the | | | | | | | | | | | | | |
| Steering Committee and the three Workgroups | | | | | | | | | | | | | |

| | <br> | <br> | _ |
|---|---|---|---|
| Obtain MOU with the KAH, and establish DMSB | | | |
| Submit data access requests to: HHS for OASIS database and to KAH for access to DEMA-Pro care plan and LMS data bases | | | |
| Identify pilot sites and DEMA Program interveners, Review/adapt HHS EHR policies and procedures. | | | |
| Refine DEMA in-person training delivery to blended learning models for DEMA-Pro | | | |
| Pilot test DEMA-Pro training and revise as needed | | | |
| Access and analyze process and outcome data from OASIS and KAH DEMA-Pro care plan and LMS databases | | | |
| Extract, link and verify accuracy of data | | | |
| Assess value of and ease of obtain outcomes measures for use in R33 | | | |

Note: IRB = Institutional Review Board; MOU = Memoranda of Understanding; HHS = Home Health Services; EHR= Electronic Health Record; DSMB = Data Safety and Monitoring Board; OASIS = Outcome and Assessment Information Set; LMS = Learning Management System; DEMA-Pro = Daily Engagement Meaningful Activity Professional